CLINICAL TRIAL: NCT05593146
Title: A Multi-center, Double-blinded, Randomized Controlled Study Comparing Modified Cup Anteversion vs Conventional Cup Anteversion Placement in Prevention of Postoperative Dislocation in Patients Undergoing Acetabular Tumor Resection and Reconstruction
Brief Title: A Randomized Controlled Study Evaluating Modified Cup Anteversion Placement in Prevention of Postoperative Dislocation in Patients Undergoing Acetabular Tumor Resection and Reconstruction
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022_QH1020
Record Dates: First submitted 2022-10-21; First posted 2022-10-25 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-01

CONDITIONS: Periacetabular Tumor
Keywords: dislocation, endoprosthetic reconstruction, anteversion angle, pelvis
MeSH Terms: conditions — Joint Dislocations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified anteversion angle placement (( α-15°)±10°) of the acetabular component (Experimental): α refers to the anatomical preoperative anteversion angle of the affected hip. α equals to the anteversion angle of the contralateral limb if it cannot be accurately measured on the affected limb. A standard error within 10° is accepted
  Interventions: Behavioral: modified anteversion angle placement(( α-15°)±10°)
- conventional anteversion angle placement ( α±10°) of the acetabular component (Placebo Comparator): α refers to the anatomical preoperative anteversion angle of the affected hip. α equals to the anteversion angle of the contralateral limb if it cannot be accurately measured on the affected limb. A standard error within 10° is accepted
  Interventions: Behavioral: conventional anteversion angle placement ( α±10°)

INTERVENTIONS:
Behavioral: modified anteversion angle placement(( α-15°)±10°) — Preoperative examination was conducted to determine a safe surgical margin in all patients. A 3D printed osteotomy guide combined with a 3D printed prosthesis pre- designed anteversion angle is assembled for reconstruction after tumor resection.
  Once completed, intraoperative X-ray fluoroscopy was applied to evaluate the anteversion angle of the acetabular component. If the anteversion angle doesn't meet the predetermined criteria, it needs to be adjusted until it does.
  Arms: modified anteversion angle placement (( α-15°)±10°) of the acetabular component
Behavioral: conventional anteversion angle placement ( α±10°) — Preoperative examination was conducted to determine a safe surgical margin in all patients. A 3D printed osteotomy guide combined with a 3D printed prosthesis with predesigned anteversion angle is assembled for reconstruction following tumor resection.
  Once completed, intraoperative X-ray fluoroscopy was applied to evaluate the anteversion angle of the acetabular component. If the anteversion angle doesn't meet the predetermined criteria, it needs to be adjusted until it does.
  Arms: conventional anteversion angle placement ( α±10°) of the acetabular component

SUMMARY:
The purpose of this clinical study is to investigate whether patients who receive modified anteversion angle (( α-15°)±10°) of the acetabular cup have a lower risk of dislocation within one year after surgery, compared to patients who receive conventional anteversion angle ( α±10°) of the acetabular cup.

The hypothesis is that patients with placement of the modified (( α-15°)±10°) anteversion angle of the acetabular component will have decreased risk of dislocation 1 year after surgery compared to patients with conventional anteversion angle ( α±10°) placement.

PS: α refers to the preoperative anteversion angle of the affected hip. α equals to the anteversion angle of the contralateral limb if it cannot be accurately measured on the affected limb. A standard error within 10° is accepted

DETAILED DESCRIPTION:
Hip dislocation is a common complication in patients who undergo reconstruction surgery after periacetabular tumor resection and most of these cases are anterior dislocations. Studies suggest that this type of dislocation may be closely related to the position and anteversion angle of the acetabular component. Therefore, properly reducing the anteversion angle of the acetabular cup during reconstruction might effectively prevent possible collisions between the cup and the femoral component, thereby reducing the potential risk of dislocation. Based on this theory, we aim to investigate whether patients who receive modified anteversion angle (( α-15°)±10°) of the acetabular cup have a lower risk of dislocation within one year after surgery, compared to patients who receive conventional anteversion angle ( α±10°) of the acetabular cup.

PS: α refers to the preoperative anteversion angle of the affected hip. α equals to the anteversion angle of the contralateral limb if it cannot be accurately measured on the affected size. A standard error within 10° is accepted.

ELIGIBILITY:
Inclusion Criteria:

* Age above 16 years old, gender is not limited.
* Tumor involving periacetabulum, femoral head, femoral neck or proximal femur
* Patients require 3D-printed hemipelvic endoprosthetic reconstruction following periacetabular tumor resection
* The subject has an estimated survival period of at least one year or more.
* The subjects with informed consent

Exclusion Criteria:

* The patient used to conduct surgery on his/her hip joint
* The patient's current surgery aimed for hip revision for implant failure or infection
* The patient didn't conduct hip endoprosthetic reconstruction
* Patients with congenital defects in the gluteal muscle group, neurological function or pelvic tilt deformity severe enough to affect functional activity
* Patients cannot self-assess postoperative function after surgery
* According to the judgment of the investigator/supervisor, there may be difficulties in completing postoperative follow-up
* Subjects have participated in similar research projects

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
The endpoint for patient participation will dislocate | followed for 1 years postoperatively for study end points
  postoperative hip dislocation

SECONDARY OUTCOMES:
MSTS score | followed 1 month, 3 months, 6 months, 9 months and 1 year postoperatively for study endpoints
  The Musculoskeletal Tumor Society (MSTS) scoring system is a validated and well-accepted functional scoring system used in orthopaedic oncology research
TESS score | followed 1 month, 3 months, 6 months, 9 months and 1 year postoperatively for study endpoints
  Toronto Extremity Salvage Score (TESS) is a physical disability measure developed specifically for patients undergoing surgery for extremity tumours
Henderson's failure mode | followed 1 month, 3 months, 6 months, 9 months and 1 year postoperatively for study endpoints
  1: soft tissue failure; 2: aseptic loosening; 3: structural failure; 4: periprosthetic infection; 5: tumor progression

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo No.6 Hospital, Ningbo, Zhejiang, China